CLINICAL TRIAL: NCT02709460
Title: Lateral Versus Cervical Coagulation of the Uterine Artery in Benign Hysterectomy: A Randomized Controlled Study
Brief Title: Lateral Occlusion of Uterine Artery in Total Laparoscopic Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Vibeke Lysdal, Consultant, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20140104
Record Dates: First submitted 2016-03-04; First posted 2016-03-16 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Postoperative Hemorrhage
Keywords: hematoma; complication; hysterectomy
MeSH Terms: conditions — Postoperative Hemorrhage; Hematoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lateral occlusion (Experimental): Women included in this arm is randomized to lateral occlusion of the uterine artery
  Interventions: Procedure: Lateral occlusion
- cervical occlusion (Active Comparator): Women included in this arm is randomized to occlusion of the uterine artery at cervical entry
  Interventions: Procedure: Cervical occlusion

INTERVENTIONS:
Procedure: Lateral occlusion — Lateral occlusion close to the internal Iliac artery
  Arms: Lateral occlusion
Procedure: Cervical occlusion — Cervical occlusion of the uterine artery
  Arms: cervical occlusion

SUMMARY:
Laparoscopic hysterectomy is associated with complications in form of infections and subsequently dehiscence of the vault. This is a serious complication. The infection may be related to the frequently observed postoperative hematoma following traditional laparoscopic hysterectomy where the uterine artery is coagulated and divided at the cervical entry into the uterus.

By coagulation of the uterine artery laterally close to the internal iliac artery this problem may be eliminated due to the much less bleeding observed during this procedure.

DETAILED DESCRIPTION:
Laparoscopic hysterectomy (removal of the uterus) is today a well-described method for the removal of the uterus. The operation is offered in case of bleeding disorders where other treatments have been unsuccessful, uterine fibroids or other conditions requiring surgery with removal of the uterus.

The operation is done today in most cases by dividing the uterine artery at the entrance to the cervix, where the artery divides into one ascending and descending branch.

The most common complication of hysterectomy is bleeding perioperative well as postoperatively, which may result in a hematoma above the vaginal vault.

Through the years different methods have been tried to reduce this complication, including tranexamic acid without great success. The hematoma may result in infection postoperative and subsequent poor healing, with the possibility of dehiscence of the vault.

In the worst case, the gut is displaced through the vagina postoperatively. This condition can lead to diffuse peritonitis, which can be fatal in rare cases.

Since the hemostasis related to the dividing of the artery uterine can be problematic, especially in case of fibroids it may be a technical advantage to coagulate the Uterine artery at the exit of the Internal Iliac artery. This operation also ensures identification of the ureter, which can be spared. Lesions to the ureter are detected in up to 1% of all surgical procedures at hysterectomy.

Dividing of the Uterine artery at the Internal Iliac Artery also ensures that the artery can be divided with minimal bleeding at the cervix.

ELIGIBILITY:
Inclusion Criteria:

* Women submitted to total laparoscopic hysterectomy

Exclusion Criteria:

* Women <18 years
* Women no able to understand the study or not native in Danish
* Women with uterine malignancy
* Women with suspicion of pelvic mass
* Women with abnormal coagulation
* Women receiving glucocorticoid treatment
* Women receiving anticoagulant treatment or have not followed prescription in relation to surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of postoperative hematoma | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Vibeke Lysdal, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No